CLINICAL TRIAL: NCT07210385
Title: Radiographic and Histomorphometric Assessment of Anterior Horizontal Maxillary Bone Augmentation Using Autogenous and Bovine Sticky Bone Versus Autogenous and Bovine Bone Shell Technique (Khoury): A Randomized Comparative Clinical Trial
Acronym: RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Seham Mohammed Ahmed Ahmed Salama, Faculty of Oral & Dental Medicine , Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: omfs 3-3-20; self funded (Other: Faculty of Oral & Dental Medicine, Cairo Univeristy)
Record Dates: First submitted 2025-09-30; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-07

CONDITIONS: Maxillary Augmentation in Horizontal Bone Defect
Keywords: Horizontal Bone Defects , Maxillary augmentation , sticky bone , bone shell technique , dental implants, alveolar ridge augmentation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Autogenous + Bovine Sticky Bone (Experimental): Participants in this group will undergo maxillary horizontal ridge augmentation using a mixture of autogenous bone chips and S1 Bovine Bone Graft in a 70:30 ratio, prepared as Sticky Bone in the area of the defect
  Interventions: Procedure: anterior horizontal maxillary bone augmentation using autogenous and bovine sticky bone
- Autogenous + Bovine Bone Shell Technique (Khoury) (Active Comparator): Participants in this group will undergo horizontal ridge augmentation using autogenous cortical bone plates harvested from the mandibular ramus fixed to the recipient site, with S1 Bovine Bone Graft used to fill the gap between plates and the alveolar bone.
  Interventions: Procedure: anterior horizontal maxillary bone augmentation using autogenous and bovine bone shell technique (khoury)

INTERVENTIONS:
Procedure: anterior horizontal maxillary bone augmentation using autogenous and bovine sticky bone — Participants in this group will undergo maxillary horizontal ridge augmentation using a mixture of autogenous bone chips and S1 Bovine Bone Graft in a 70:30 ratio. The graft will be prepared as Sticky Bone and applied to the defect site for augmentation.
  Arms: Autogenous + Bovine Sticky Bone
Procedure: anterior horizontal maxillary bone augmentation using autogenous and bovine bone shell technique (khoury) — Participants in this group will undergo maxillary horizontal ridge augmentation using the Khoury Bone Shell Technique, combining autogenous bone blocks and Bovine Bone Graft to reconstruct the alveolar ridge. The graft will be fixed and stabilized to provide a rigid shell for bone regeneration.
  Arms: Autogenous + Bovine Bone Shell Technique (Khoury)

SUMMARY:
This clinical trial aims to compare two bone augmentation techniques for patients with anterior horizontal maxillary bone defects:

Autogenous and Bovine Sticky Bone Technique using S1 Bovine Bone Graft Autogenous and Bovine Bone Shell Technique (Khoury Technique). The study will evaluate the amount of bone gain and the quality of bone formation after six months using radiographic (CBCT) and histomorphometric analysis. Patients will be randomly assigned to one of the two groups and followed for six months post-surgery to assess bone regeneration, surgical outcomes, and potential complications.

DETAILED DESCRIPTION:
This randomized controlled clinical trial will be conducted at the Department of Oral and Maxillofacial Surgery, Faculty of Oral and Dental Medicine, Cairo University. The study addresses the clinical challenge of horizontal maxillary bone defects, which complicate implant placement and require effective augmentation techniques.

Two techniques will be compared:

Autogenous and Bovine Sticky Bone: Using S1 Bovine Bone Graft mixed with autogenous bone chips in a 70:30 ratio.

Autogenous and Bovine Bone Shell Technique (Khoury): Using autogenous cortical bone shells harvested from the mandible combined with S1 Bovine Bone.

The primary outcome is horizontal bone gain assessed by CBCT immediately after surgery and at six months before implant placement. Secondary outcomes include histomorphometric analysis of bone core biopsies to evaluate the quality of bone regeneration.

Randomization will be performed with a 1:1 allocation ratio using computer-generated sequences. Patients will be blinded to the intervention, and follow-up will be conducted at 3 days, 1 week, 1 month, 2 months, and 6 months postoperatively.

The trial aims to determine whether the less invasive sticky bone technique can achieve comparable or superior bone regeneration outcomes compared to the traditional bone shell method while reducing donor site morbidity and surgical complexity

ELIGIBILITY:
Inclusion Criteria

* Patients aged 18-55 years.
* Both males and females.
* Patients with horizontal bone deficiency in the anterior maxillary region (< 3 mm width) requiring augmentation prior to implant placement.
* Adequate oral hygiene and commitment to follow-up visits.

Exclusion Criteria:

* Patients with systemic diseases affecting bone healing (e.g., uncontrolled diabetes, osteoporosis).
* Heavy smokers (>10 cigarettes/day).
* Pregnant or lactating women.
* Previous bone grafting procedures at the same site.
* Patients on medications affecting bone metabolism (e.g., bisphosphonates).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-01-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Anterior Horizontal Maxillary Alveolar ridge bone gain | Baseline (immediately post-surgery) 6 months after augmentation
  The primary outcome measure will be the amount of horizontal bone gain at the augmented site measured in millimeters using Cone Beam Computed Tomography (CBCT). Measurements will be taken immediately after augmentation and at 6 months before implant placement.

SECONDARY OUTCOMES:
Quality of bone formation | Up to 6 months
  Bone core biopsy will be obtained at the time of implant placement to assess the percentage of newly formed bone, residual graft material, and connective tissue using histomorphometric analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Al Manyal, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share individual participant data (IPD) has not yet been made. Data sharing will depend on institutional review board (IRB) approvals, institutional policies, and participant consent. If data sharing is approved in the future, detailed information about the process, access conditions, and timelines will be provided.

REFERENCES:
- [Background] Shaker AE, Salem AS, El-Farag SA, Abdel-Rahman FH, El-Kenawy MH. Comparison of Khoury's Bone Shell Technique vs Titanium-reinforced Polytetrafluoroethylene Membrane for 3D-bone Augmentation in Atrophic Posterior Mandible: A Randomized Clinical Trial. J Contemp Dent Pract. 2024 Jun 1;25(6):518-526. doi: 10.5005/jp-journals-10024-3704. PMID 39364817
- [Background] Tony JB, Parthasarathy H, Tadepalli A, Ponnaiyan D, Alamoudi A, Kamil MA, Alzahrani KJ, Alsharif KF, Halawani IF, Alnfiai MM, Ramachandran L, Balaji TM, Patil S. CBCT Evaluation of Sticky Bone in Horizontal Ridge Augmentation with and without Collagen Membrane-A Randomized Parallel Arm Clinical Trial. J Funct Biomater. 2022 Oct 19;13(4):194. doi: 10.3390/jfb13040194. PMID 36278663
- [Background] Yazhini P K, Suresh N, Kaarthikeyan G. Subperiosteal Ridge Augmentation Technique Utilizing Sticky Bone: A Case Series. Cureus. 2024 Jul 29;16(7):e65641. doi: 10.7759/cureus.65641. eCollection 2024 Jul. PMID 39205712
- [Background] Barbu HM, Iancu SA, Rapani A, Stacchi C. Guided Bone Regeneration with Concentrated Growth Factor Enriched Bone Graft Matrix (Sticky Bone) vs. Bone-Shell Technique in Horizontal Ridge Augmentation: A Retrospective Study. J Clin Med. 2021 Aug 31;10(17):3953. doi: 10.3390/jcm10173953. PMID 34501399
- [Background] De Angelis P, Cavalcanti C, Manicone PF, Liguori MG, Rella E, De Rosa G, Palmieri A, D'Addona A. A Comparison of Guided Bone Regeneration vs. the Shell Technique Using Xenogeneic Bone Blocks in Horizontal Bone Defects: A Randomized Clinical Trial. Dent J (Basel). 2024 May 9;12(5):137. doi: 10.3390/dj12050137. PMID 38786535